CLINICAL TRIAL: NCT03121443
Title: The Association Between Surgical Patient Positions and Perfusion Index
Brief Title: Patient Positions and Perfusion Index
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 17-KAEK-2017
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-05

CONDITIONS: Perfusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient position: Perfusion index
  Interventions: Other: Perfusion index

INTERVENTIONS:
Other: Perfusion index — supine,prone, trendelenburg,reverse trendelenburg,45 degrees back up sitting position, 45 degrees legs lifted supine position.

SUMMARY:
The association between patient positions including supine,prone, trendelenburg,reverse trendelenburg,45 degrees back up sitting position, 45 degrees legs lifted supine position and perfusion index.

DETAILED DESCRIPTION:
Participants are taken to the recovery room and they will wait 15 minutes until measurements. After monitoring the perfusion index using the right ring finger, first the participant will be taken to supine position. The perfusion index value will be obtained after three minutes of measurement. Second, the position will change to 45 degrees back up sitting position and the measurement will be repeated. Then the participant will be taken to Trendelenburg position, reverse Trendelenburg position, prone, 45 degrees legs lifted supine position respectively, and same measurement will perform.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists score of 1

Exclusion Criteria:

* any kind of disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers American society of anesthesiologists score of 1
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-07-02 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Perfusion index | one month
  Perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Principal Investigator — Assistan professor
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No